CLINICAL TRIAL: NCT01675388
Title: Hypothermia as Neuroprotection During ECMO: Is Brain MRI a Biomarker of Outcomes?
Brief Title: Hypothermia During ECMO to Decrease Brain Injury
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding
Sponsor: Sood, Beena G., MD, MS (Individual)
Responsible Party: Principal Investigator, Beena G. Sood, MD, MS, Associate Professor, Sood, Beena G., MD, MS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1006008466
Record Dates: First submitted 2012-08-24; First posted 2012-08-30 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Neonatal Respiratory Failure
Keywords: Neonatal hypoxemic respiratory failure; Extra Corporeal Membrane Oxygenation; Neurodevelopmental outcomes; Neuroimaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hypothermia (Experimental): Hypothermia to 33.5 deg Centigrade
  Interventions: Other: Hypothermia

INTERVENTIONS:
Other: Hypothermia — Hypothermia to 33.5 deg C

SUMMARY:
Newborn infants with severe respiratory failure are treated with extracorporeal membrane oxygenation (ECMO), a modified form of cardiopulmonary bypass. These infants as at risk for brain injury as a result of hypoxia and blood flow changes in the brain prior to and during ECMO. The investigators propose a clinical trial of a novel treatment (cooling during ECMO) and novel diagnostic tool (advanced MRI techniques) that will lead to improved outcomes, early diagnosis and intervention for brain injury, decreased cost and duration of clinical trials, decrease in the burden of chronic neurologic disease and disability in society, thus improving the health and quality of life of these infants as they progress through childhood into adulthood.

DETAILED DESCRIPTION:
Term and late preterm neonates with severe hypoxemic respiratory failure [NHRF] receive extracorporeal membrane oxygenation (ECMO), a modified form of cardiopulmonary bypass, when maximal conventional therapy fails. Although ECMO significantly improves survival and decreases disability, 15-50% of survivors nevertheless have poor neurodevelopmental [ND] outcomes due to hypoxemia and cerebral hypoperfusion occurring prior to and during ECMO. Hypothermia [HYP] (33 deg-34 deg C for 48-72 hours) has been shown to improve ND outcomes and following neonatal hypoxic-ischemic encephalopathy [NE]. Whether the addition of hypothermia to ECMO for severe NHRF will improve ND outcomes is unknown. Long-term evaluation of ND outcomes is the gold standard for determining the full spectrum of developmental disabilities as neonatal clinical findings; biochemical and electrophysiological tests; and cranial sonography have limited predictive value. Conventional magnetic resonance imaging [MRI] has a predictive accuracy of > 0.8 for death and disability following NE. MR abnormalities in infants undergoing ECMO for NHRF differ from those seen in NE and there are no systematic reports on the ND implications of MR abnormalities seen in NHRF treated with ECMO. Given the societal and economic costs associated with poor long-term ND outcomes and the challenges of neurologic assessment in critically ill neonates receiving ECMO for NHRF, there is an urgent need for (i) neuroprotection pre-/during ECMO to decrease brain injury and (ii) innovative diagnostic modalities to enable early diagnosis and intervention.

Our goal is to improve the treatment and ND outcomes in neonates with NHRF. The overall objectives of this proposal are to establish the neuroprotective role of hypothermia during ECMO for NHRF as evaluated by ND assessment at 18-22 months [mo] of age and to validate the use of conventional and advanced MR techniques as biomarkers of brain injury. The central hypotheses are that (i) HYP to 33.5°C during the 1st 72 hours of ECMO in NHRF will reduce the extent and severity of brain injury as evaluated by Bayley Scales of Infant Development (BSID-III) cognitive scores at 18-22 mo and proportion of normal MRI studies in the neonatal period and at 18-22 mo; and (ii) conventional and advanced MR techniques in the neonatal period and at 18-22 mo will be biomarkers of brain injury allowing prediction of ND outcomes, and monitoring of post-injury brain growth and plasticity.

The specific aims are to evaluate:

1. Safety and efficacy of hypothermia combined with ECMO for NHRF in improving neurodevelopmental outcomes at 18-22 months of age
2. MR abnormalities in the neonatal period and at 18-22 months of age and their predictive accuracy for neurodevelopmental outcomes at 18-22 months of age following hypothermia during ECMO for NHRF

MRI will be obtained in the neonatal period as part of routine clinical care; MRI will be repeated at 18-22 mo of age on an outpatient basis if funding is available to assess longitudinal changes in brain structure and metabolite profile following ECMO for NHRF and to correlate these with ND outcomes at 18-22 mo of age.

ELIGIBILITY:
Inclusion Criteria:

* Neonates ≥ 34 weeks gestational age and postnatal age ≤ 28 days
* Presence of severe reversible NHRF qualifying for ECMO based on institutional guidelines including:

  * Oxygenation Index > 35 ([mean airway pressure in cmH2O x Fractional inspired O2 concentration x 100]/Arterial O2 tension in mmHg) or
  * Alveolar-arterial oxygen gradient > 600 mmHg for 4 h
* Infants undergoing veno-arterial or veno-venous ECMO

Exclusion Criteria:

* Lethal chromosomal and congenital anomalies including congenital diaphragmatic hernia (CDH) Infants with CDH, who constitute a third of neonates undergoing ECMO, have been excluded because the high mortality and morbidity is related more to the underlying lung abnormality and practice variation in timing of CDH repair rather than to NHRF.
* ECMO for post operative cardiac support
* Neonates with a birth weight < 1.8 kg
* Initiation of HYP for NE prior to initiating ECMO for NHRF

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
BSID-III cognitive scores at 18-22 mo | 18-22 months of age

SECONDARY OUTCOMES:
Clinical findings in the neonatal period and at 18-22 mos | 18-22 months
  i) outcomes in the neonatal intensive care unit (NICU): HUS findings, type of ECMO, death/withdrawal of intensive care, acute AEs, cardio-respiratory support, infections, need for gavage/gastrostomy-tube feeds, length of hospital stay, bronchopulmonary dysplasia, neurologic status, and growth parameter at discharge ii) outcomes after discharge: post-neonatal deaths, number of re-hospitalizations, seizure disorder, growth parameters, BSID-III subscales at 18-22 mo, visual impairment, hearing impairment, multiple disabilities
MRI findings in the neonatal period and at 18-22 mos | 18-22 months
  MRIs at 18-22 months will only be evaluated if funding for obatining MRIs becomes available

CONTACTS AND LOCATIONS:
Overall Officials: Beena G. Sood, Principal Investigator — Wayne State University
Locations (1):
- Children's Hospital of Michigan, Detroit, Michigan, United States